CLINICAL TRIAL: NCT05734300
Title: Organ SPARring Surgery vs. Standard Resection for Early Stage COLon Cancer in Elderly Frail Patients
Brief Title: The "SPARCOL" Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EMN 2022-04791
Record Dates: First submitted 2023-01-16; First posted 2023-02-17 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Colon Cancer; Frailty
Keywords: Colon Cancer; Elderly population; Early colo-rectal cancer; Organ Preserving Approach; Combined Endoscopic Laparoscopic Surgery (CELS)
MeSH Terms: conditions — Colonic Neoplasms; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CELS (Experimental): The Combined Endoscopic Laparoscopic Surgery (CELS) is a hybrid procedure that enables large local excisions of the colon without segmental resection while under general anaesthesia. In our study, CELS refers only to endoscopic assisted laparoscopic resection.
  Interventions: Procedure: Combined Endoscopic Laparoscopic Surgery (CELS)
- Standard Surgery (Active Comparator): Standard surgical resection of colonic cancer following standard oncologic principles while under general anaesthesia.
  Interventions: Procedure: Standard resection

INTERVENTIONS:
Procedure: Combined Endoscopic Laparoscopic Surgery (CELS) — The main surgical advantage in this procedure is the ability to view the colon intra- and extraluminal simultaneously. The laparoscopic approach enables manipulation and mobilization of the colon, while the endoscopic view secures that the resection is complete and not overlapping the ileac valve or creating stenosis.
  Compared to the traditional oncological colon resection, the CELS resection is a minimally invasive procedure - organ sparing procedure leading to a reduced surgical stress response.
  Arms: CELS
Procedure: Standard resection — In this study standard resection of the colon will be performed according to complete mesocolic excision (CME) principles.
  Arms: Standard Surgery

SUMMARY:
Mortality following elective colorectal cancer surgery range between 2.5-6% and increase for the elderly and frail patient regardless of T-stage. Around 80% of the patients who present with a colon cancer and is in a condition where surgery is possible will be offered resection of the tumor. A part of the colon is always removed together with the lymph nodes in order to ensure that cancer cells are not left behind. The risk of lymph node metastasis is dependent on several histopathological characteristics of the tumor. The overall risk of lymph node metastases is less than 20 % in patients with early colon cancer. This indicates that the majority of patients with early colon cancer have no benefit of additional resection besides local tumor excision. The alternative to resecting a larger part of the bowel is to make more focused surgery only resecting a small part of the bowel part through a combination of laparoscopic and endoscopic techniques. This new organ sparing approach is called Combined Endoscopic Laparoscopic Surgery (CELS). The investigators aimed to examinate the hypothesis that organ preserving approach (CELS) provides superior quality of recovery in elderly frail patients with small colon cancers when compared with standard surgery in RCT.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female participants providing written informed consent aged 75 years and older
* PS score ≥1 and /or ASA score ≥3
* Macroscopically or pathological colonic adenocarcinoma
* Clinical TNM classification T1/T2 N0 M0
* Eligible and suitable for CELS resection according to MDT
* Tumor must be located in colon, and not involving the ileac valve or taking up more than 50% of the lumen in an air-distended bowel wall

Exclusion Criteria:

* Unable to give informed consent
* Histological high-risk features in biopsy material from tumor (mucin, signet cells, de- differentiation)
* Suspected other malignancy than adenocarcinoma (e.g. neuroendocrine tumors)
* Preoperative chemo/radiotherapy
* Creation of stoma perioperative
* Non-Danish speakers

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in patient-reported postoperative recovery - Quality of Recovery 15 | Change in QoR-15 will be assessed repeatedly at baseline, 4-8 hours postoperatively (4-8H), postoperative day (POD) 1, POD 2, POD 3, POD 7, POD 10-14 and POD 30
  Validated to measure recovery after surgery and general anesthesia, and additionally validated for use in Danish language and culture. The scale is arbitrary and ranges from 0 to 150. Higher scores means better recovery. The established minimum clinically important difference in QoR-15 is 8.0, and the SD of QoR- 15 scores after major surgery is in the order of 16.

SECONDARY OUTCOMES:
Change in exercise capacity and physical condition | Changes will be assessed repeatedly at baseline, Postoperative day 1, Postoperative day 2, Postoperative day 3 or at the time of hospital discharge, whatever comes first. Postoperative day 10-14 and 30 days postoperatively.
  The 30 Second Sit to Stand Test. A measurement that assesses functional lower extremity strength in older adults. Test result is the number of times the participant comes to a full standing position in 30 seconds. Higher number of stands within 30 seconds means better result.
Change in exercise capacity and physical condition | Changes will be assessed repeatedly at baseline, Postoperative day 1, Postoperative day 2, Postoperative day 3 or at the time of hospital discharge, whatever comes first. Postoperative day 10-14 and 30 days postoperatively.
  Six minutes' walk test is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes.
Changes in The European Organization for Research and Treatment of Cancer quality of life questionnaire - EORTC C30. | Changes will be assessed repeatedly at basline, 3 months, 6 months, 1 year follow-up
  EORTC C30, questionnaire, developed to assess the quality of life of cancer patients. All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the patient).
Changes in The European Organization for Research and Treatment of Cancer quality of life questionnaire- EORTC CRC. | Changes will be assessed repeatedly at basline, 3 months, 6 months, 1 year follow-up
  EORTC CRC questionnaire, developed to assess the quality of life of cancer patients. All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the patient).
Frailty questionnaire Geriatric 8 (G8) | Basline
  The G-8 Score is a screening tool containing 8 questions. The total G-8 score lies between 0 and 17. A higher score indicates a better health status.
Duration of surgery | Intraoperative
  Duration of surgery in minutes
Blood loss | Intraoperative
  Blood loss in ml
Intraoperative complications | Intraoperative
  Descriptive registration of intraoperative complications;
Conversion rate | Intraoperative
  Conversion rate (%) from laparoscopic surgery to open surgery
Rate of complete resection margin | Postoperative day 14
  R0 (tumor-free margin >1 mm) corresponds to resection for cure or complete remission. R1 to microscopic residual tumor, R2 to macroscopic residual tumor.
Assessment of histopathological risk factors | Postoperative day 14
  Assessment of histopathological risk factor defined as presence of at least one of the risk factors: Kikuchi level ≥sm2, vascular invasion, lymphatic invasion, poorly differentiated adenocarcinoma, and tumour budding BD2-3.
Long-term oncological outcomes: Disease-free survival | During 3-year follow-up periode
  Time from surgery until the recurrence of disease or death
Long-term oncological outcomes: Overall survival | During 3-year follow-up periode
  Overall survival was defined as the time elapsed from the date of surgery to the last day of follow-up or the date of death
Long-term oncological outcomes: Recurrence | During 3-year follow-up periode
  Locoregional and/or distant recurrence after surgery defined as any histological, morphological, and clinical evidence of tumour growth during follow-up periode
Clavien-Dindo classification | Within 90 days postoperative.
  Grading system used in surgery for grading adverse events (i.e. complications) which occur as a result of surgical procedures. Grade I to V, where V is death of the patient
The Comprehensive Complication Index | Within 90 days postoperative.
  e Comprehensive Complication Index (CCI®) reflects the gravity of this overall complication burden on the patient on a scale from 0 (no complication) to 100 (death)
Length of hospital stay | Within 90 days postoperative.
  Clinical metric that measures the length of time in days elapsed between a patient's hospital admittance and discharge.
90-day mortality | Within 90 days postoperative.
  Death within 90 days after surgery, as either an inpatient or outpatient
Hospital readmissions | Within 90 days postoperative.
  Unplanned readmissions that happen within 3 days of discharge from the index (i.e., initial) admission
Rate of secondary standard resection | Within 90 days postoperative.
  Rate in percent of performed secondary surgery after primary CELS resection

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Copenhagen University Hospital - Herlev, Copenhagen, Herlev
  - Hospital Soenderjylland, Aabenraa
  - Zealand University Hospital, Køge